CLINICAL TRIAL: NCT03032692
Title: Motor Task Performance Under Visual and Auditory Feedback Post Stroke: a Randomized Crossover Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Collaborators: CMM - Centro Médico da Murtosa (Unknown); CMM - Centro Médico de Aveiro (Unknown); Centro Médico de Viseu (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RCT-BFK01
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Stroke; Upper Extremity Paresis
MeSH Terms: conditions — Ischemic Stroke; Paresis | interventions — Exercise; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SWORD and exercise with biofeedback (Experimental): The patient will perform one repetition of the exercise shoulder flexion with elbow flexion at 90 degrees under monitoring from SWORD. The recorded parameters will be used to define: baseline and target angle; execution time; maximum postural sway. Two additional repetitions will be performed to ensure reproducibility. During the session, SWORD will be providing real-time audiovisual feedback. The patient has to start in the baseline position and fill the progress bar without violating movement or posture constraints. If the patient does not reach the goal or violates constraints he will receive a negative audio feedback, the progress bar will turn red and be reset. The patient has to return to the baseline position to restart the movement.
  Interventions: Device: SWORD; Other: Exercise with biofeedback
- SWORD and exercise without biofeedback (Active Comparator): The patient will perform one repetition of the exercise shoulder flexion with elbow flexion at 90 degrees under monitoring from SWORD. The recorded parameters will be used to define: baseline and target angle; execution time; maximum postural sway. Two additional repetitions will be performed to ensure reproducibility. The patient will then be instructed to perform as many movements as possible during the allocated time (4 minutes), at a comfortable pace, starting at or below the baseline and trying to reach maximum flexion without significant pain or discomfort. During the session, the SWORD system will be recording the patient´s movement without providing feedback to the patient.
  Interventions: Device: SWORD; Other: exercise without biofeedback

INTERVENTIONS:
Device: SWORD — Both arms will perform two separate sessions consisting of one exercise - shoulder flexion with elbow flexion at 90 degrees - for 4 minutes in two experimental conditions: with and without biofeedback. Group 1 will perform the exercise with biofeedback first and without biofeedback after; group 2 performed the exercise in the opposite order. The SWORD system will be used to record movement data in both sessions.
  Other Names: Stroke Wearable Operative Rehabilitation Device
Other: Exercise with biofeedback
  Arms: SWORD and exercise with biofeedback
Other: exercise without biofeedback
  Arms: SWORD and exercise without biofeedback

SUMMARY:
The study was designed to evaluate the impact of a novel kinematic biofeedback system - SWORD - in the motor performance of patients after stroke. The SWORD system combines inertial motion trackers and a mobile app, allowing digitization of patient motion and providing real-time audiovisual biofeedback.

The investigators hypothesize that the biofeedback feedback provided by the SWORD system improves patient performance, defined as an increase in the number of correct movements.

The design of the study is a cross-over randomized clinical trial. Patients will be randomized into two groups. Both will perform two separate sessions consisting of one exercise - shoulder flexion with elbow flexion at 90 degrees - for 4 minutes in both experimental settings: with and without biofeedback. Group 1 will perform the exercise with biofeedback first and without biofeedback after, with an interval >24h. Group 2 will perform the exercise in the opposite order. The SWORD system will be used to record movement data in both sessions, but the feedback was only active in one of them.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms and signs and CT or MRI findings compatible with a lesion in the territory of the medial cerebral artery;
* persistent motor deficit on the upper limb but not plegia with a score between 0 and 2 on item 5b of the National Institute of Health Stroke Scale (NIHSS)
* more than 2 weeks after stroke onset;
* the ability to sit comfortably for more than 10 minutes and perform two-step commands

Exclusion Criteria:

* no detectable motor deficits at baseline assessment;
* severe aphasia;
* clinical dementia or mini mental state examination (MMSE) below cutoff;
* other cognitive or psychiatric comorbidity that impaired communication or compliance with the tasks;
* severe respiratory or cardiac condition incompatible with more than 5 minutes of continuous mild exercise in a sitting position;
* pain or deformity that limited upper limb movement on the affected side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Number of correct movements | At the end of each exercise session (4 minute duration)
  Number of correct movements performed within the duration of each exercise session

SECONDARY OUTCOMES:
Total number of repetitions | At the end of each exercise session (4 minute duration)
  Total number of repetitions performed within the duration of each exercise session
Number of incorrect repetitions | At the end of each exercise session (4 minute duration)
  Number of incorrect repetitions performed within the duration of each exercise session
Number of consecutive incorrect repetitions | At the end of each exercise session (4 minute duration)
  Number of consecutive incorrect repetitions performed within the duration of each exercise session
Number of pauses | At the end of each exercise session (4 minute duration)
  Number of pauses registered during each exercise session
Posture errors | At the end of each exercise session (4 minute duration)
  Number of posture errors registered during each exercise session
Movement frequency | At the end of each exercise session (4 minute duration)
  Movement frequency (in Hertz) during each exercise session
Range of motion of correct movements | At the end of each exercise session (4 minute duration)
  Mean range of motion of the correct movements performed during each exercise session
Range of motion variability over time | Between the second and first minute; between the second and third minutes; between the third and fourth minute
  Variability of the mean range of motion during the exercise session (for correct movements)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — Sword Health, SA
Locations (3):
- Portugal (3):
  - CMM - Murtosa, Murtosa, Aveiro District
  - CMM - Centro Médico de Aveiro, Aveiro
  - CMM- Centro Médico de Viseu, Viseu

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be made available to other researchers